CLINICAL TRIAL: NCT00026533
Title: Phase II Trial of Thalidomide for Therapy of Radioiodine-Unresponsive Papillary and Follicular Thyroid Carcinomas and Medullary Thyroid Carcinomas
Brief Title: Thalidomide in Treating Patients With Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Ain (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kenneth Ain, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Purpose: Treatment
Other Study IDs: CDR0000069053; UKMC-IRB-010069
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV papillary thyroid cancer; stage IV follicular thyroid cancer; thyroid gland medullary carcinoma; recurrent thyroid cancer; insular thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Carcinoma, Medullary; Thyroid Neoplasms | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of thyroid cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness thalidomide in treating patients who have thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of thalidomide, in terms of tumor response and duration of response, in patients with metastatic follicular, papillary, or medullary thyroid carcinoma that is unresponsive to systemic radioiodine.
* Compare the differences in antitumor activity of this drug in patients with medullary carcinomas vs those with papillary or follicular carcinomas.
* Determine the toxic effects and duration of toxic effects of this drug in these patients.

OUTLINE: Patients receive oral thalidomide once daily for 2 weeks and then twice daily. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular, papillary, insular, or medullary thyroid carcinoma
* Must meet criteria for 1 of the following:

  * Unresectable, distantly metastatic tumor that does not concentrate radioactive iodine
  * Follicular or papillary thyroid carcinoma with a large distant tumor burden that has not sufficiently responded to cumulative iodine I 131 doses exceeding 800 mCi
* Radiographic evidence of tumor progression, meeting 1 of the following criteria:

  * Evidence gathered over a period of at least 1 year with at least 3 separate x-ray studies, defining tumor volume
  * Similar radiographic evidence over a shorter period of time, delineating more than 30% increase in tumor volume

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 750/mm^3
* Hemoglobin at least 10.5 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN
* BUN no greater than 1.5 times ULN

Other:

* No active infection not controlled with medications
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double contraception (1 hormonal method plus 1 barrier method OR 2 simultaneous barrier methods) for female patients or barrier contraception for male patients for more than 4 weeks prior to, during, and for at least 4 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior thalidomide
* No other concurrent biologic therapy

Chemotherapy:

* At least 4 weeks since prior systemic chemotherapy
* No concurrent systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed
* Concurrent limited external-beam radiotherapy to isolated sites of bony metastases allowed, provided that these sites are not the sole sites of metastatic disease and do not constitute the sites of evaluable disease for this study
* No concurrent radioiodine therapy

Surgery:

* See Disease Characteristics
* Prior surgery allowed
* Concurrent surgery allowed to sites that do not constitute evaluable disease for this study

Other:

* No concurrent medications that are known to increase the risk of peripheral neuropathy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2003-11 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ain, MD, Study Chair — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky, United States